CLINICAL TRIAL: NCT01509222
Title: Changing Dietary Patterns: an Individually Tailored Nutrition Intervention
Brief Title: Changing Dietary Patterns: an Individually Tailored Nutrition Intervention (OKE-study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Lisette de Groot, (Hooft van Huysduynen), Wageningen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL36582.081.11
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Health promotion; Dietary Counseling
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized nurition counseling (Other): Personalized nutrition counseling based on dietary intake and motivation to change.
  Interventions: Behavioral: Personalized nutrition counseling
- Control (No Intervention): No intervention, control group.

INTERVENTIONS:
Behavioral: Personalized nutrition counseling
  Arms: Personalized nurition counseling

SUMMARY:
The main objective of this study is to investigate the effect of a personalized nutrition intervention on the dietary pattern of apparently healthy adults with one or more children aged 4 to 12 years.

DETAILED DESCRIPTION:
Giving personalized nutrition advice is perceived to be more effective in changing dietary patterns than giving general information about healthy eating.

ELIGIBILITY:
Inclusion Criteria:

* At least aged 18 years
* Having one child aged 4 to 12 years
* Written informed concent has been obtained

Exclusion Criteria:

* Not meeting the inclusion criteria
* Unable or unwilling to comply with the study procedures
* Enrolled in another study during the same study period
* Not being able to communicate (read, speak and write) in the Dutch language
* Having a partner who has been enrolled in the study
* Being pregnant or lactating during the study period or planning to become pregnant during the study period
* Having a BMI lower than 18.5 or higher that 35 kg/m2
* Using medication to lower cholesterol or being under control by a doctor for having too high cholesterol levels
* Using medication to lower blood pressure or being under control by a doctor for having a high blood pressure.
* Having diabetes type I or type II
* Following a diet (medical or self-initiated) or planning to follow a diet during the study period
* Undergoing a medical treatment that interferes with the intervention.
* Having gained or lost more than 5 kg of body weight during the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in dietary pattern | baseline and 6 months
  Dietary pattern will be measured by scoring several aspects of the diet. There are 10 aspets included in the score; fruit consumption, vegetable consumption, fiber intake, fatty acids intake, trans fatty acids intake, physical activity, consumption occasions, alcohol intake, fish consumption and sodium intake.
  The range of the score is from 0 to 100. The score will be based on the information of a Food Frequency Questionnaire and two 24 hour dietary recalls.

SECONDARY OUTCOMES:
Dietary behaviour | baseline and 6 months
  Behavioral factors influencing dietary intake like barriers for having a healthy diet.
Health outcomes | baseline and 6 months
  Health outcome measure are; BMI, waist and hip circumference, blood lipids (cholesterol and triglycerides) and blood pressure
Markers of intake | baseline and 6 months
  Blood values of carotenoids and fish fatty acids will be used to assess whether measured changes in dietary pattern are also found in the blood.
  Urinary potassium and sodium ratios will also be used to assess changes in dietary pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne HM De Vries, Dr., Principal Investigator — Departement Human Nutrition, Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands